CLINICAL TRIAL: NCT06667479
Title: Effects of a 4 Week Cold Tub Vs Cold Shower Immersion Intervention on Immune Function, Sleep Quality, Mental Health and Well-being, Gut Health, and Muscular Strength in Healthy, Physically Active Adults
Brief Title: Cold Water Exposure and Immune Function Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2404058883
Record Dates: First submitted 2024-10-10; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Cold Water Immersion; Immune Function; Muscular Strength; Mental Health
Keywords: Cold Water Immersion; Cold Tub; Cold Shower; Immune Function; Mental Health; Muscular Strength; Healthy Adults; Inflammation; Gut Health
MeSH Terms: conditions — Psychological Well-Being; Inflammation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel, randomized design, matched for biological age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cold Tub Immersion Group (CI) (Experimental): Participants will utilize the research cold tub (10 ºC, 4-minutes, 3 times a week), following a standardized protocol (see intervention description).
  Interventions: Other: Cold Water Immersion (CWI) - Cold Tub Immersion (CI)
- Cold Shower Group (CS) (Experimental): Participants will utilize the research shower area (10 ºC, 4-minutes, 3 times a week), following a standardized protocol (see intervention description).
  Interventions: Other: Cold Water Immersion (CWI) - Cold Shower (CS)
- Control Group (CO) (Other): Participants will not undergo any cold tub or cold shower intervention.
  Interventions: Other: Control Group (CO)

INTERVENTIONS:
Other: Cold Water Immersion (CWI) - Cold Tub Immersion (CI) — Once thermoneutral procedures are complete, participants in the CI group will be seated in the cold tub and submerged into the water (10º C). The sternal notch of each participant will be used as the anatomical marker to mark submersion point. Participants will sit with both arms outstretched underwater with their backs not touching the sides of the tub. Participants with a shorter stature will be provided an underwater cushion to meet the submersion requirements. The 4-minute timer will begin once confirmation of the participants submersion level and posture is determined. Once completed, the participant will be instructed to slowly exit the tub and allowed to dry and change as necessary.
  Arms: Cold Tub Immersion Group (CI)
Other: Cold Water Immersion (CWI) - Cold Shower (CS) — Once thermoneutral procedures are complete, participants in the CS group will be instructed to enter the research shower area. Within the shower area, the walls of the shower will be numbered from 1 to 4, with 1 defined as facing the faucet, 2 defined as 90° to the right of side 1, 3 defined as 180° from the faucet, and 4 defined as 270° to the right or 90° C to the left from side 1. Participants will be instructed to turn 90° to the right cycling through sides 1 to 4 and then back to 1 every 15 seconds prompted by the researcher. This will allow the participant to complete four full rotations in the shower during the 4-minute intervention time. The shower faucet is modified and oriented in a way where it only produces cold water (10º C) when turned on. Once completed, the participant will be instructed to slowly exit the shower and is allowed to dry and change as necessary
  Arms: Cold Shower Group (CS)
Other: Control Group (CO) — Participants will be encouraged to maintain their current diet and exercise across the duration of the 4 week intervention. Participants will still be subjected to the pre- and post-intervention data collection session.
  Arms: Control Group (CO)

SUMMARY:
The purpose of this clinical trial is to explore the effects of a 4 week cold-water immersion (CWI) intervention on measures of immune function, sleep quality, mental health and well-being, and muscular strength. The main questions it aims to answer are:

* Does a 4 week CWI intervention improve measures of immune function, sleep quality, mental health and well-being, and muscular strength?
* Are there any differences in these measures when comparing cold tubs versus cold showers?

Researchers will compare chronic use of cold tubs to cold showers to see if cold water immersion may improve overall immune health and well-being.

Participants will:

* Undergo 4 weeks of Cold Tub or Cold Shower interventions at a frequency of 3 times a week for 4 minutes, if placed in the CWI intervention groups
* Undergo testing measures at the two pre- and post- intervention time points, if placed in the healthy control group or the CWI intervention groups

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Aged 18-45

Exclusion Criteria:

* Currently practices CWI for [>3 times in the last month]
* Pregnant or planning to become pregnant
* Chronic use of anti-inflammatory medication
* Prior history of chronic disease conditions:
* Cardiovascular Disease
* Diabetes
* Cancer
* Raynaud's Disease
* Severe and untreated anxiety or depression

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 60mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-min at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of CRP will be determined with a commercially available enzyme-linked immunosorbent assay (ALPCO Diagnostics, Salem, NH, USA). Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Lipopolysaccharide Binding Protein (LBP) | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 60mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-min at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of LBP will be determined with a commercially available enzyme-linked immunosorbent assay (Abcam Limited, Cambridge, UK). Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Zonulin (Haptoglobin-2 Precursor) | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 60mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-min at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of Zonulin will be determined with a commercially available enzyme-linked immunosorbent assay (Thermo Fisher Scientific, Waltham, MA, USA). Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Interleukin-6 (IL-6) | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 60mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-min at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of IL-6 will be determined with a commercially available enzyme-linked immunosorbent assay (Thermo Fisher Scientific, Waltham, MA, USA). Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Visit 1A (Week 1) and 2A (Week 4): 10 minutes each
  Participants will be asked to complete a paper version of the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-question self-reported sleep quality tool broken up into 7 subcategories for scoring, such as subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. There are also 5 additional questions directed to the respondent's roommate or bed partner not used in the scoring, but utilized for clinical purposes.
Depression Anxiety and Stress Scales (DASS-21) | Visit 1A (Week 1) and 2A (Week 4): 10 minutes each
  Participants will be asked to complete a paper version of the 21-item Depression Anxiety and Stress Scale (DASS-21). The DASS-21 consists of 21 questions using a 0-3 Likert scale assessing the participant's subjective mental health and stress state with a "0" indicating "Did not apply to me at all" and "3" indicating "Applied to me very much or most of the time." The DASS-21 contains 3 sub scales assessing Depression, Anxiety, and Stress consisting of 7 questions for each sub scale, where a high score of 28+ indicates "Extremely Severe" levels of Depression, a high score of 20+ indicates "Extremely Severe" levels of Anxiety, and a high score of 34+ indicates "Extremely Severe" levels of Stress, while low scores of 0-9 indicates "Normal" levels of Depression, scores of 0-7 indicates "Normal" levels of Anxiety, and scores of 0-14 indicates "Normal" levels of Stress.
Handgrip Dynamometry | Visit 1B (Week 1) and Visit 2B (Week 4): 10 minutes each
  Isometric grip strength will be measured by a Baseline 12-0286 Electronic Smedly Hand Dynamometer (Fabrication Enterprises, White Plains, NY). To begin the test, participants will stand upright in a relaxed position; their upper extremity peak isometric grip strength will be assessed with the shoulder in 180º of flexion, elbow at full extension, and wrist and forearm in a neutral position. When prompted, participants will squeeze the device with their dominant hand, delivering a maximal effort for 3-seconds, followed by relaxation. After 30-seconds, the test will be run again. Three sets are completed for this test, and the highest value (kg) will be recorded for analysis.
Gastrointestinal Symptoms Questionairre (GSQ) | Completed During Visit 1A and 2A (10 minutes)
  Participants will be asked to complete an online version of the Gastrointestinal Symptoms Questionnaire (GSQ). The GSQ is a 29-question self-reported gastrointestinal (GI) screening tool broken up into two subcategories for scoring, one for their GI symptoms experienced today and the other for their GI symptoms experienced in the last 4 weeks. There are also two open-ended question at the end of the survey, one describing any other GI symptoms not addressed in the questionnaire and another addressing normal food consumption. The GSQ will be completed online during Visits 1A and 2A.

OTHER OUTCOMES:
Lean Body Mass | Visit 1A (Week 1) and Visit 2A (Week 4): 20 minutes each
  Lean body mass (LBM) will be evaluated using air displacement plethysmography using a calibrated BODPOD (COSMED USA Inc., Concord, CA). Participants will be instructed to remove their shoes, socks, jewelry, and all additional clothing other than their base layer. Participants will then be given a swim cap to wear and body composition analysis will be performed per the manufacturer's guidelines.
Body Fat Percentage | Visit 1A (Week 1) and Visit 2A (Week 4): 20 minutes each
  Body fat percentage (BF%) will be evaluated using air displacement plethysmography using a calibrated BODPOD (COSMED USA Inc., Concord, CA). Participants will be instructed to remove their shoes, socks, jewelry, and all additional clothing other than their base layer. Participants will then be given a swim cap to wear and body composition analysis will be performed per the manufacturer's guidelines.
Immune Status Questionnaire (ISQ) | Visit 1A (Week 1): 5 minutes
  Participants will be asked to complete a paper version of the Immune Status Questionnaire (ISQ). The ISQ consists of 7 items rating the respondent's past year's immune status, by inquiring about the incidence of specific immune-related complaints. The ISQ helps to establish participant's perceived immune fitness based on the previous 12 months incidence of disease symptoms. The ISQ utilizes a 0-4 Likert scale to evaluate incidence of these symptoms where a 0 indicates "Never" and a 4 indicates "Always (Almost)." The raw scores are added and converted into a final score where a final score of 0 indicates "very poor perceived immune status," while a final score of 10 indicates "excellent perceived immune status." Final scores less than 6 will be classified as reduced perceived immune function.
CWI Perceptions Qualitative Assessment | Visit 1A (Week 1) and Visit 2A (Week 4): 10 minutes each
  Participants will be asked to complete a qualitative questionnaire to indicate their perceptions of cold water therapy before and after the study. The purpose of this assessment is to see if participants' perceptions changed throughout the study. Further, this questionnaire allows participants to provide any extra qualitative feedback to gain a comprehensive insight on their chronic CWI experience. No scale is used in this survey; however, participants are given the opportunity to report their perceptions of cold immersion using the following choices: increases energy, reduces anxiety, improves sleep, improves mental health, improves physical health, improves immune system, reduces soreness or pain, or other [text response].
Visual Analogue Scale (VAS) of Discomfort | Each CWI Intervention Session: 10 seconds
  During each session of cold therapy, participants will be assessed on their subjective ratings of discomfort as they acclimate to the cold exposure. During (at 1-minute mark) cold-water immersion, participants will be presented with the Visual Analogue Scale (VAS) of Discomfort, a modified version of a 0-10 item pain scale. This version of the VAS is a subjective measure of discomfort using a 11-point Likert scale ranging from 0 - 10 with 0 indicating "No Discomfort" and 10 indicating "Maximal Discomfort."
Natural Killer Cell Count | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 8 hours.
  Approximately 15 mL venous whole blood was collected per participant in heparinized vacutainers. The samples were placed on ice and the Peripheral Blood Mononuclear Cells (PBMC) were isolated within 4 h of collection. Whole blood was mixed at a 1:1 ratio with ice cold DPBS. PBMCs were isolated by layering onto a Ficoll Paque density gradient medium, and then centrifuged at 400 xg for 40 min at 18 °C. PBMC were then washed in DPBS and resuspended in complete RPMI 1640 (10% FBS, 1% Penicillin-Streptomycin) medium at 1.0 × 106 cells/mL. PBMCs were stained with efluro450-conjugated anti-CD3 and PerCP-efluro 610-conjugated anti-CD56 (Invitrogen, Carlsbad, CA) for 20 min on ice and in the dark for expression of CD56+/CD3- NK cells and CD56+/CD3+ NKT cells. PBMCs were washed with ice cold DPBS following staining to remove excess antibody and resuspended in ice cold DPBS for analysis via flow cytometry. The percentage of NK cells were determined as a proportion of total PBMCs.
Natural Killer T Cell Count | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 8 hours.
  Approximately 15 mL venous whole blood was collected per participant in heparinized vacutainers. The samples were placed on ice and the Peripheral Blood Mononuclear Cells (PBMC) were isolated within 4 h of collection. Whole blood was mixed at a 1:1 ratio with ice cold DPBS. PBMCs were isolated by layering onto a Ficoll Paque density gradient medium, and then centrifuged at 400 xg for 40 min at 18 °C. PBMC were then washed in DPBS and resuspended in complete RPMI 1640 (10% FBS, 1% Penicillin-Streptomycin) medium at 1.0 × 106 cells/mL. PBMCs were stained with efluro450-conjugated anti-CD3 and PerCP-efluro 610-conjugated anti-CD56 (Invitrogen, Carlsbad, CA) for 20 min on ice and in the dark for expression of CD56+/CD3- NK cells and CD56+/CD3+ NKT cells. PBMCs were washed with ice cold DPBS following staining to remove excess antibody and resuspended in ice cold DPBS for analysis via flow cytometry. The percentage of NK T cells were determined as a proportion of total PBMCs.
Natural Killer Cell Cytotoxicity Assay | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 8 hours.
  Chronic human myelogenous leukemia cells (K562; ATCC, Manassas, VA) were used to evaluate NK cell effector function. K562 cells were stained with Alexa-Fluro 647-conjugated anti-CD71. K562 cells were further stained with Calcein-AM viability dye (Thermo Fisher Scientific, Waltham, MA) on ice and in the dark for 20 min. K562 cells were washed and resuspended at 1.0 × 106 cells/mL in complete RPMI 1640 medium. Human PBMCs containing effector NK and NKT cells were co-cultured with target K562 cells in 5 mL eppendorf tubes at a 40:1 PBMC:K562 effector: target (E:T) ratio and incubated for 4 h at 37 °C in a cell incubator. Following co-incubation, samples were centrifuged at 400 xg for 5 min and resuspended in ice cold DPBS for analysis. After the 4-hour co-culture, these samples were analyzed via flow cytometry to determine the total proportion of alive (Calcein-AM+) versus dead (SYTOX Blue+) K562 cells.Changes in proportion and MFI of these populations were further analyzed using FlowJo.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Northern Colorado - Gunter Hall, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All study documents will be made available upon reasonable request (Laura.stewart@unco.edu).
Time Frame: Oct 1, 2025 - Oct 1, 2028
Access Criteria: Individuals will email Laura.stewart@unco.edu with a request for study materials.